CLINICAL TRIAL: NCT01208896
Title: Safety and Efficacy of a Strategy of Allogeneic Hematopoietic Stem Cell Transplantation After Reduced-intensity Conditioning for Chemosensitive Relapsed Follicular Lymphoma
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation After Reduced-intensity Conditioning for Relapsed Follicular Lymphoma
Acronym: RITALLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/09
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Follicular; Stem Cell Transplantation
Keywords: Allogeneic hematopoietic stem cell transplantation; Reduced-intensity conditioning; Chemosensitive relapsed follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Reduced_intensity conditioning

INTERVENTIONS:
Drug: Reduced_intensity conditioning — The conditioning regimen is composed of Fludarabine (30 mg/m2) and Cyclophosphamide (750 mg/m2), both administered intravenously at Days -5, -4, -3 with Day 0 being the day of transplantation. Rituximab will be administered intravenously at 375 mg/m2 at Day -13 and 1000 mg/m2 at Days -6, +1, +8. Tacrolimus and low-doses of methotrexate will be used for prophylaxis of GVHD.

SUMMARY:
This trial will evaluate the efficacy and the safety of a strategy of allogeneic stem cell transplantation including Rituximab in the conditioning regimen for the treatment of relapsed follicular lymphoma. The rationale for using Rituximab relies on a better control of the disease and a better prophylaxis of the graft versus host disease.

DETAILED DESCRIPTION:
Follicular lymphomas are chemosensitive neoplasms characterized by a relentless succession of remissions and relapses when treated with conventional chemotherapy. The successive periods of remission are of shorter duration and patients invariably die of their disease. At first line, patients are treated with conventional chemotherapy. At first relapse, intensive chemotherapy with autologous stem cell transplantation (SCT) is often proposed.

Allogeneic hematopoietic stem cell transplantation after reduced-intensity conditioning (RIC-allo) is an option for patients relapsing after autologous SCT, allowing long-term progression free survival of 50 to 60%. The toxic mortality related to severe acute graft versus host disease (GVHD) remains a critical issue. The goal of our study is to test in a multicentric approach a strategy of RIC-allo including rituximab in order to reduce the incidence of acute GVHD.

Around half of patients with relapsed or refractory follicular lymphomas treated with allogeneic SCT achieve long-term progression free survival whatever the conditioning regimen. Because the median age of patients with follicular lymphoma is 55 years, a reduced intensity conditioning is the most appropriate option in this setting. The outcome of patients with a chemoresistant disease is usually poor because of a high toxic mortality. As a consequence, only patients with a chemosensitive disease will be included in this study. To further reduce the toxic mortality, it is critical to reduce the incidence of severe acute GVHD. A low incidence of acute GVHD could be obtained by the use of Rituximab before and after the transplantation as reported by the MD Anderson's experience in several hematological malignancies including follicular lymphoma. Their results are impressive in patients with follicular lymphoma with long-term survival of 85%. The favored hypothesis is a depletion of patient and donor B cells reducing the presentation of minor histocompatibility alloantigens. The benefit of Rituximab could also be explained by its anti-lymphoma effects that could compensate the putative reduction of a graft versus lymphoma effect due to a better control of GVHD.

The primary objective is to estimate 2-year overall survival in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years
* Follicular lymphoma confirmed by a biopsy at the last relapse.
* 2nd, 3rd or 4th complete or partial response according to Cheson's criteria 1 (Annexe 1)
* Relapse after autologous-SCT except if the absence of autologous SCT is due to a failure of collecting peripheral stem cells or investigator decision to not proceed to the autologous graft because of serious criteria
* Relapse after at least one line of treatment with rituximab
* Karnofsky index > 70%
* HLA Matched related or unrelated donor (10/10 matching; HLA-A, HLA-B, HLA-C, HLA-DRB1, HLA-DQB1)
* Signed informed consent

Exclusion Criteria:

* Stable or progressive disease according to Cheson's criteria1 (Annexe 1)
* Absence of treatment with rituximab before the last relapse
* Cardiac insufficiency (ejection fraction < 50% by echocardiography)
* Pulmonary disease characterized by DLCO < 60%
* Renal insufficiency (clearance of creatinin < 60 ml/min)
* Hepatic disease characterized by ASAT and/or ALAT and/or total bilirubin > 2 times the upper normal value except in case of Gilbert's disease or hepatic lymphoma
* HIV positive test
* Bacterial, Viral or Fungal uncontrolled infections
* Pregnant or breast feeding woman
* Cancer in the last 5 years except in case of cutaneous baso-cellular cancer or epithelioma "in situ" of the uterine cervix

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-02-03 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 year

SECONDARY OUTCOMES:
Toxic mortality | 2 year
Progression free survival | 2 year
Incidence of relapse | 2 year
Grade II-IV acute GVHD incidence | 2 year
Chronic GVHD incidence | 2 year
Morbidity and adverse event | 2 year
Hematologic reconstitution, Immunologic reconstitution, Chimerism | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane VIGOUROUX, MD, Principal Investigator — University Hospital, Bordeaux
Locations (26):
- France (26):
  - University Hospital Angers, Angers, Angers
  - Service Hématologie, Hôpital Minjoz, Besançon
  - Service Hématologie, Hôpital Augustin Morvan, Brest
  - University Hospital, Caen, Caen
  - Service Hématologie et Thérapie cellulaire, Pavillon Villemin Pasteur, CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Service Hématologie Oncologie, Hôpital Lapeyronie, CHU de Montpellier, Montpellier
  - CHU Nancy, Nancy
  - Service Hématologie Clinique, CHU -Hôtel Dieu, Nantes
  - Service Hématologie Clinique, Hôpital Archet 1, Nice
  - APHP Hôpital Necker-Enfants malades, Paris
  - APHP Hôpital Saint Louis, Paris
  - APHP Hôpital Pitié-Salpêtrière, Paris
  - APHP Hôpital Henri-Mondor, Paris
  - Service des maladies du sang - Hôpital Haut-Lévêque - avenue de magellan, Pessac
  - CHU Poitiers - La Milétrie, Poitiers
  - Service Hématologie Clinique, Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - Département d'Hématologie et d'Oncologie, Hôpital CHRU de Hautepierre, Strasbourg
  - Service Hématologie, Hôpital Purpan, Toulouse
  - CHRU Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Khouri IF, Saliba RM, Giralt SA, Lee MS, Okoroji GJ, Hagemeister FB, Korbling M, Younes A, Ippoliti C, Gajewski JL, McLaughlin P, Anderlini P, Donato ML, Cabanillas FF, Champlin RE. Nonablative allogeneic hematopoietic transplantation as adoptive immunotherapy for indolent lymphoma: low incidence of toxicity, acute graft-versus-host disease, and treatment-related mortality. Blood. 2001 Dec 15;98(13):3595-9. doi: 10.1182/blood.v98.13.3595. PMID 11739162
- [Background] Khouri IF, McLaughlin P, Saliba RM, Hosing C, Korbling M, Lee MS, Medeiros LJ, Fayad L, Samaniego F, Alousi A, Anderlini P, Couriel D, de Lima M, Giralt S, Neelapu SS, Ueno NT, Samuels BI, Hagemeister F, Kwak LW, Champlin RE. Eight-year experience with allogeneic stem cell transplantation for relapsed follicular lymphoma after nonmyeloablative conditioning with fludarabine, cyclophosphamide, and rituximab. Blood. 2008 Jun 15;111(12):5530-6. doi: 10.1182/blood-2008-01-136242. Epub 2008 Apr 14. PMID 18411419
- [Background] Vigouroux S, Michallet M, Porcher R, Attal M, Ades L, Bernard M, Blaise D, Tabrizi R, Garban F, Cassuto JP, Chevalier P, Facon T, Ifrah N, Renaud M, Tilly H, Vernant JP, Kuentz M, Bourhis JH, Bordigoni P, Deconinck E, Lioure B, Socie G, Milpied N; French Society of Bone Marrow Graft Transplantation and Cellular Therapy (SFGM-TC). Long-term outcomes after reduced-intensity conditioning allogeneic stem cell transplantation for low-grade lymphoma: a survey by the French Society of Bone Marrow Graft Transplantation and Cellular Therapy (SFGM-TC). Haematologica. 2007 May;92(5):627-34. doi: 10.3324/haematol.10924. PMID 17488686
- [Background] Christopeit M, Schutte V, Theurich S, Weber T, Grothe W, Behre G. Rituximab reduces the incidence of acute graft-versus-host disease. Blood. 2009 Mar 26;113(13):3130-1. doi: 10.1182/blood-2009-01-200527. No abstract available. PMID 19324911